CLINICAL TRIAL: NCT03530865
Title: Assessment of the Variations in the Number of Roots and the Root Canal System of the Permanent Mandibular First and Second Molars in a Sample of Egyptian Population Using Cone Beam Computed Tomography
Brief Title: Assessment of the Variations in the Root Canal System of the Permanent Mandibular First and Second Molars Among Egyptian Population Using Cone Beam Computed Tomography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farid Medhat, Principal Investigator, Cairo University
Other Study IDs: RAD2:8:7
Record Dates: First submitted 2018-04-02; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Number of Roots; Number of Root Canals
Keywords: mandibular molars; extra root; extra root canal; root morphology; cbct endodontics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study to estimate Variations in the Number of Roots and the Root Canal System of the Permanent Mandibular First and Second Molars in a Sample of Egyptian Population using cone beam computed tomography through retrospective data analysis

DETAILED DESCRIPTION:
Setting and Location:

The data collection will be obtained from the data base available at the department of oral and maxillofacial radiology, faculty of dentistry, Cairo university, Cairo, Egypt.

cone beam images will be obtained from Egyptian patients who had cone beam computed tomography examination as part of their dental examination, diagnosis or treatment planning .

Participants:

A total sample of 384 mandibular first and second permanent molars belonging to Egyptian individuals will be included.

Images of the first and second mandibular permanent molars are selected according to the following criteria:

Inclusion criteria:

* Fully maturated and erupted mandibular permanent first and second molars of Egyptian patients, males or females .
* Intact roots without fractures or cracks .
* Molars without posts or previous root canal treatment .
* cone beam scans of mandibular first and second molars using different fields of view, and different voxel resolutions .

Exclusion criteria:

* Evidence of apicectomy or periapical surgery .
* Mandibular molars with developmental anomalies .
* External or Internal Root resorption .
* Root Canal Calcification .
* Previous Root Canal treatment .
* Post restorations .
* Root caries specially reaching the bifurcation area .
* Tomographic images of poor quality or artifacts interfering with the detection of root canals .

Variables:

1. Number of roots of mandibular first and second molars .
2. Number of root canals of mandibular first and second molars .

Data Sources / Measurements:

* Retrospective Data Analysis will be performed after the Cone beam images are pooled from the computer database.
* All the cone beam computed tomography examinations will be scanned using CBCT Software (Planmeca Romexis Viewer) .
* cone beam computed tomography images will be analysed in the 3 planes; first the sagittal and coronal sections will be oriented parallel to the long axis of the root, and then sections will be obtained on the axial plane for detection of the number of roots and root canals.
* cone beam computed tomography images will be interpreted by three oral radiologists independently; blinded from demographic data of the patients and from the results of each other.
* Each one will evaluate the images separately twice with a period of two weeks between the two reading sessions.
* Then inter-observational and intra-observational variability between the observers will be evaluated.

Bias:

No source of bias.

Study Size:

To detect variations in number of roots and root canals in permanent mandibular first and second molars in the Egyptian population. The investigators are going to apply convenient consecutive sampling.Using a precision of 5, a design effect set at 1 with 95% CI (confidence interval), a total sample size of 384 will be sufficient. The sample size was calculated by Epi info.

sampling strategy: The sample will be collected by simple random sampling .

Quantitative Variables:

The number of cone beam computed tomography scans of Egyptian individuals with extra roots and accessory root canals in mandibular first and second permanent molars will be counted to estimate the variations in the Egyptian population.

Statistical methods:

Data will be analysed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 21 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages. Comparisons between male and females for normally distributed numeric variables will be done using the Student's t-test while for non-normally distributed numeric variables will be done by Mann-Whitney test. Comparisons between categorical variables will be performed using the chi square test. A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.

ELIGIBILITY:
Inclusion Criteria:

* Fully maturated and erupted mandibular permanent first and second molars of Egyptian patients, males or females .
* Intact roots without fractures or cracks .
* Molars without posts or previous root canal treatment .
* CBCT scans of mandibular first and second molars using different fields of view, and different voxel resolutions .

Exclusion Criteria:

* Evidence of apicectomy or periapical surgery .
* Mandibular molars with developmental anomalies .
* External or Internal Root resorption .
* Root Canal Calcification .
* Previous Root Canal treatment .
* Post restorations .

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian population
Sampling Method: Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Extra root in the first and second mandibular permanent molars | six months
  by Percentage

SECONDARY OUTCOMES:
Extra root canals in the first and second mandibular permanent molars | six months
  by percentage